CLINICAL TRIAL: NCT06467513
Title: To Investigate the Effect of Esketamine on Hemodynamics and Postoperative Pulmonary Complications in Patients Undergoing Heart Valve Replacement Surgery
Brief Title: To Investigate the Effect of Esketamine Hydrochloride on Pulmonary Complications
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Zhang XIao Mei (Other)
Responsible Party: Sponsor-Investigator, Zhang XIao Mei, Anesthesiology resident, Affiliated Hospital of Zunyi Medical University, Zunyi Medical College
Organization: Zunyi Medical College (Other)
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Other
Other Study IDs: KLL-2023-223
Record Dates: First submitted 2024-06-14; First posted 2024-06-21 (Actual); Last update posted 2024-06-21 (Actual); Status verified 2024-06

CONDITIONS: Heart Diseases; Heart Valve Diseases
MeSH Terms: conditions — Heart Diseases; Heart Valve Diseases | interventions — Sodium Chloride

STUDY DESIGN:
Intervention Model Description: This study was divided into 3 groups, one group was placebo group, the other group was low-dose esketamine group (continuous injection of esketamine until the end of surgery), the dose was 0.2mg/kg; The other group was the Esketamine high-dose group (the continuous injection of esketamine during the operation until the end of the operation) with a dose of 0.4mg/kg.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The randomized personnel of the study enrolled suitable patients according to the random number table method before surgery, and then extracted drugs for anesthesia (anesthesia and patients did not know the group). The group status was not known to the post-operative follow-up personnel or the data analysts.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- blank control group (No Intervention): In the blank control group, no intervention was used during the operation, and normal saline was pumped according to the participant's body weight until the end of the operation.
- Low dose esketamine hydrochloride injection group (Experimental): In the low-dose ESketamine hydrochloride injection group, 50mg of Esketamine hydrochloride injection was diluted with normal saline into a 50ml syringe, which was wrapped with light-proof paper and pumped continuously from the beginning of anesthesia to the end of surgery. The dosage was calculated as 0.2mg/kg.h.
  Interventions: Drug: Esketamine hydrochloride injection
- High dose esketamine hydrochloride injection group (Experimental): In the high-dose ESketamine hydrochloride injection group, 50mg of Esketamine hydrochloride injection was diluted with normal saline into a 50ml syringe, which was wrapped with light-resistant paper and pumped continuously from the beginning of anesthesia to the end of surgery. Dosage was calculated as 0.4mg/kg.h.
  Interventions: Drug: Esketamine hydrochloride injection

INTERVENTIONS:
Drug: Esketamine hydrochloride injection — The low dose esketamine hydrochloride group was given 0.2mg/kg at induction of anesthesia, the high dose esketamine hydrochloride group was given 0.4mg/kg at induction of anesthesia, and the blank control group was not given Esketamine hydrochloride injection at induction of anesthesia.
  Other Names: 0.9% sodium chloride injection
  Arms: High dose esketamine hydrochloride injection group; Low dose esketamine hydrochloride injection group

SUMMARY:
The objective of this study was to evaluate the effect of esketamine on intraoperative hemodynamics in patients with heart valve replacement and to mitigate postoperative pulmonary complications

DETAILED DESCRIPTION:
After being informed of the study and potential risks, all patients who gave written informed consent will undergo pre-operative screening to determine eligibility for study enrollment. Before operation, eligible patients were randomly divided into esketamine group (0.2mg/kg, intraoperative pump), esketamine group (0.4mg/kg, intraoperative pump) and blank control group (physiological salt pump) in a double-blind way at a ratio of 1:1:1.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-75 years old, gender unlimited.
* Elective heart surgery.
* Patients who plan to undergo mitral and (or) aortic valve replacement (or repair) surgery, requiring extracorporeal circulation and aortic occlusion.
* The New York Heart Association class is less than 4.
* Voluntarily sign informed consent.

Exclusion Criteria:

* Non-cardiac surgery.
* Second heart surgery.
* Interventional surgery in heart valve surgery (TAVI, mitral clamp).
* The patient refuses.
* Pregnant women.
* Patients with a history of lung surgery.
* Patients with acute kidney injury requiring dialysis.
* Patients with chronic renal insufficiency (stage III and above).
* The patient was intubated before arriving at the operating room.
* Patients with existing pulmonary complications (respiratory tract infection, pneumonia, pleural effusion, respiratory failure, atelectasis, pneumothorax, bronchospasm, ARDS).
* The patient had neuropsychiatric disease and cognitive impairment before surgery.
* Drug users and other long-term use of antipsychotic drugs.
* Patients with any of the following contraindications for the use of ESketamine injection: patients with serious risk of elevated blood pressure or intracranial pressure; Patients with high intraocular pressure (glaucoma) or penetrating ocular trauma; Patients with poorly controlled or untreated hypertension (arterial hypertension, resting systolic pressure exceeding 180 mmHg, or resting diastolic pressure exceeding 100mmHg); Patients with untreated or undertreated hyperthyroidism (hyperthyroidism).
* Liver function ALT, AST > 2 times normal.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Pulmonary ultrasound score | Baseline and day 1, day 2 and day 3 after surgery
  The anterior axillary line, posterior axillary line and paraspinal line were used as the boundary, and each lung was divided into 3 regions: anterior chest, underarm and back. Each area was given a maximum score of 3 out of 36, with higher scores indicating worse lung condition.

SECONDARY OUTCOMES:
The concentration of interleukin 6 | At baseline, before anesthesia induction, 10 minutes after insertion of tracheal catheter, 10 minutes after cardiopulmonary bypass, 10 minutes after completion of cardiopulmonary bypass, at the end of surgery, and 1 day after completion of surgery.
  The concentration of interleukin-6 in participants before and during surgery, as well as after surgery, can reflect the size of the inflammatory response to some extent.

CONTACTS AND LOCATIONS:
Overall Officials: Wei Chen, Study Director — Staff member of Department of Anesthesiology, Affiliated Hospital of Zunyi Medical University; Haiying Wang, Principal Investigator — Director of anesthesiology Department, Affiliated Hospital of Zunyi Medical University
Locations (1):
- Affiliated Hospital of Zunyi Medical University, Zunyi, Guizhou, China

IPD SHARING:
Plan to Share IPD: Yes
After the clinical trial, each subgroup and its corresponding lung ultrasound score were shared with other research teams.
Supporting Information: CSR
Time Frame: Data related to this trial can be shared for a total of 6 months after publication.
Access Criteria: Contact the head of the study for approval